CLINICAL TRIAL: NCT06049342
Title: A Phase I, Open Label, Single Arm, Multiple Center, Dose Escalation Clinical Trial to Evaluate the Safety, Tolerability and Efficacy of Human Induced Pluripotent Stem Cell Derived Mesenchymal Stromal Cells (NCR100) Injection in the Treatment of Subjects With Knee Osteoarthritis
Brief Title: A Trial to Evaluate the Safety, Tolerability, and Efficacy of NCR100 Injection in the Treatment of Subjects With KOA
Acronym: NCR100
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nuwacell Biotechnologies Co., Ltd. (Industry)
Collaborators: Shanghai 6th People's Hospital (Other); Beijing Luhe Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCR100-1001
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Knee Osteoarthritis
Keywords: KOA; Mesenchymal Stromal Cells
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NCR100 injection (Experimental): Cohort1:Low dose NCR100 injection; Cohort2:Mid-low dose NCR100 injection; Cohort3:Mid-high dose NCR100 injection; Cohort4:High dose NCR100 injection.
  Interventions: Biological: NCR100 injection

INTERVENTIONS:
Biological: NCR100 injection — Subjects will receive a one-dose intra-articular NCR100 injection.

SUMMARY:
This clinical study is to investigate the safety and efficacy of NCR100 injection in subjects with knee osteoarthritis (KOA). It is a dose-escalating, open label study in adult KOA subjects.

DETAILED DESCRIPTION:
Knee osteoarthritis (KOA) is a kind of degenerative joint disease and there are over 300 million cases worldwide. The aim of this clinical trial is to evaluate the safety, tolerability, and efficacy of human pluripotent stem cell derived mesenchymal stromal cells (NCR100) injection in the treatment of subjects with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who understand and voluntarily sign the Informed Consent Form（ICF） before the enrolment;
* Age: 40-80 years old, both genders;
* Diagnosis of knee osteoarthritis based on American College of Rheumatology criteria;
* Subjects with KOA who have persistent pain for more than six months, or aggravation or recurrence of osteoarthritis after routine medication;
* Kellgren-Lawrence grade: II-III;
* McMaster Universities Osteoarthritis Index (WOMAC): 24-72.

Exclusion Criteria:

* Subjects previously diagnosed of secondary knee osteoarthritis, or those diagnosed with hip/ankle joint disease requiring medical intervention;
* Subjects who suffering from other diseases that cause damage to knee joint function or affect joints;
* Subjects who have received allogeneic mesenchymal progenitor (stem/stromal) cell therapy;
* Subjects who have history of knee joint injury;
* Subjects who have undergone knee arthroscopic surgery;
* Subjects who received painkillers ( eg,opioids/nonsteroidal anti-inflammatory analgesics ) to treat knee osteoarthritis;
* Subjects who have orally taken traditional Chinese medicine;
* Subjects who have received intra-articular drug injection to treat knee osteoarthritis;
* Subjects with glucosamine, chondroitin sulfate, or diacetate therapy before investigational drug intervention
* Subjects with acute reactive knee osteoarthritis;
* Severe eversion deformity in target knee joint;
* Known or suspected allergy or a history of allergies;
* Subjects with abnormal results of laboratory examination: Hepatic Insufficiency (ALT > 2xULN or Aspartate aminotransferase（AST） > 2xULN), renal dysfunction (creatinine clearance rate ≤60ml/min or blood urea nitrogen(BUN) > 2× ULN), Coagulation Defects (INR > 1.5) or severe hematological diseases (Grade 3 or above anemia Hb < 8 g/dL, Grade 2 or above thrombocytopenia platelet count(PLT) < 75×10^9/L) ;
* BMI≥30 kg/m^2 ;
* Severe systemic infection or local knee joint infection;
* Subjects who have received systemic glucocorticoid therapy before intervention or need to take systemic glucocorticoid therapy during the treatment;
* Subjects who have history of acute myocardial infarction or with heart diseases e.g.uncontrolled angina pectoris, uncontrolled arrhythmias, severe heart failure (NYHA > III), QT prolongation, and are determined by investigators as not suitable to participate in this clinical trial;
* Subjects with peripheral or central nervous system disorders that may interfere with knee joint pain and functional assessment,
* Subjects who have contraindications to MRI;
* Subjects who have poor physical condition and are unable to walk autonomously;
* Subjects with alcohol or drug addiction or with a clear history of mental disorders or with a history of drug abuse or drug use of psychotropic substances;
* Subjects with infection with hepatitis B virus(HBV), hepatitis C virus(HCV), HIV, and treponema pallidum confirmed by laboratory tests;
* Pregnant or lactating female subjects, or subjects who are unable to comply with contraceptives from the study period to 6 months after the end of this study;
* Subjects who have participated in other clinical trials and have used other study products;
* Subjects with severe and poorly controlled comorbidities and not suitable for this clinical trial;
* Subjects who are not suitable for this clinical trial for other reasons.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-01-25 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Adverse Event(AE) or Serious Adverse Event(SAE) | Week1,Week2,Week4
  Number of participants with treatment-related adverse events or serious adverse events as assessed by CTCAE v5.0
Dose-Limiting Toxicity(DLT) | 4 weeks after injection
  Number of participants with Dose-limiting toxicity in 28 days after injection

SECONDARY OUTCOMES:
Maximum plasma concentration(Cmax) | 30minutes before administration,24hours,1week,2week,4week,8week,12week and 24week after administration
Elimination half life of drug(T1/2) | 30minutes before administration,24hours,1week,2week,4week,8week,12week and 24week after administration
Time after doing at which maximun plasma concentration is reached(Tmax) | 30minutes before administration,24hours,1week,2week,4week,8week,12week and 24week after administration
Area under the plasma concentration-time curve(AUC) | 30minutes before administration,24hours,1week,2week,4week,8week,12week and 24week after administration

CONTACTS AND LOCATIONS:
Overall Officials: Changqing Zhang, Principal Investigator — Shanghai 6th People's Hospital

IPD SHARING:
Plan to Share IPD: No